CLINICAL TRIAL: NCT04891653
Title: A Open-label, Multi-center Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics and Efficacy of BR790 Monotherapy in Subjects With Advanced Solid Tumors
Brief Title: A Phase I Study of BR790 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QF-BR790-101
Record Dates: First submitted 2021-05-11; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5-65mg QD (Experimental)
  Interventions: Drug: BR790

INTERVENTIONS:
Drug: BR790 — Subjects will receive oral administration of BR790.

SUMMARY:
The purpose of the study was to evaluate the safety and tolerability of BR790 tablets as an oral monotherapy in subjects with advanced solid tumors, and to determine dose-limiting toxicity (DLT), maximum tolerated dose (MTD) and/or recommended phase II clinical trial dose (RP2D) .The study is divided into two phases: dose escalation phase and dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent voluntarily.
* Age ≥18 and ≤75 years old.
* Subjects with advanced solid tumors diagnosed by histology or cytology，whose desease progressed after standard treatment or have no standard treatment.
* Had at least one measurable lesion.
* ECOG≤1.
* Expected survival period ≥ 3 months.

Exclusion Criteria:

* Any previous treatment with SHP-2 inhibitor.
* Symptomatic brain metastases.
* Subjects with thoracic/ascites fluid that need drainage or intervention.
* Subjects with not enough organ functional reserve at baseline, which met at least one of the following criteria： ANC<1.5×10^9/L PLT<100×10^9/L Hb<90g/L TBIL>1.5×ULN ALT, AST>2.5×ULN (without liver metastases) or ALT, AST>5×ULN (with liver metastases), Cr >1.5×ULN.
* With uncontrolled severe disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | up to 32 day
maximum tolerated dose (MTD) | up to 32 day
recommended phase II clinical study dose (RP2D) | up to 32 day

SECONDARY OUTCOMES:
AUC | up to 32 day
Cmax | up to 32 day
t1/2 | up to 32 day
pERK | up to 32 day
  the level of pERK in blood
AE | through study completion, an average of 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
ORR | through study completion, an average of 3 years